CLINICAL TRIAL: NCT07362407
Title: Analysis of the Therapeutic and Clinical Profile of Cannabinoid Treatments: A Real-World Study (CANAREAL)
Brief Title: Analysis of the Therapeutic and Clinical Profile of Cannabinoid Treatments: A Real-World Study
Acronym: CANAREAL
Status: Not yet recruiting | Type: Observational
Sponsor: Santa Catarina Federal University (Other)
Collaborators: HempMeds Brasil (Unknown)
Responsible Party: Principal Investigator, Taynara da Silva, Master's Degree, Santa Catarina Federal University
Other Study IDs: CANAREAL-2025; 8.083.335 (Other: Ethics Committee in Research of the Federal University of Santa Catarina)
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Depression Disorders; Anxiety Disorders; Quality of Life; Cannabidiol Effects; Cannabinoids
Keywords: cannabis; cannabinoids; medical cannabis; Real-Word Evidence; Quality of life; observational study; cbd; thc; brazil; chronic pain
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders; Marijuana Abuse; Color Vision Defects; Wiskott-Aldrich Syndrome | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Medicinal Cannabinoid Users: Patients who use or are starting treatment with cannabis-based products prescribed under Brazilian regulations (RDC 660/22). This group includes individuals seeking treatment for various clinical conditions, such as chronic pain, anxiety, and depression, through compassionate use.
  Interventions: Other: Participants are followed while using cannabis-based products (such as CBD or THC oils, extracts, or isolates) as prescribed by their own physicians for therapeutic purposes.

INTERVENTIONS:
Other: Participants are followed while using cannabis-based products (such as CBD or THC oils, extracts, or isolates) as prescribed by their own physicians for therapeutic purposes. — This is an observational study of patients using cannabis-based products as prescribed by their personal physicians. The investigators do not provide, prescribe, or assign any medication. Participants will use various formulations (such as CBD-dominant, THC-dominant, or balanced full-spectrum oils) administered according to their specific medical guidance. Data collection will focus on the natural course of the treatment, monitoring clinical evolution, quality of life, and safety through validated scales over a 6-month period.
  Other Names: Cannabis-based products; Phytocannabinoids; CBD oil; medical marijuana; Full-spectrum

SUMMARY:
What is the purpose of this study? The use of medicinal cannabis has grown significantly in Brazil. However, because many patients use these products through "compassionate use" (when traditional treatments haven't worked), there is still a lack of large-scale data on how these treatments perform in daily life. This study, called CANAREAL, aims to track patients across Brazil to understand if cannabis-based products are truly effective and safe for treating various conditions, such as chronic pain, anxiety, and depression.

How will the study work? This is an observational study, which means the researchers will not provide the medication or change the treatment prescribed by the patient's doctor. Instead, we will simply "follow" the patient's journey for 6 months.

What will participants be asked to do? Participants will complete online questionnaires at different stages of their treatment. These tools will measure:

Quality of Life: How the treatment affects daily well-being.

Clinical Evolution: Changes in pain levels, anxiety, and depression symptoms.

Safety: Whether the patient experiences any side effects (adverse events).

Why is this study important? Unlike controlled laboratory tests, this "Real-World Study" captures the reality of diverse patients with different backgrounds and health needs. The information gathered will help doctors, patients, and health authorities in Brazil better understand the benefits and risks of cannabinoid therapy, leading to safer and more informed medical decisions in the future.

DETAILED DESCRIPTION:
Study Rationale and Context The CANAREAL study is designed as a prospective, longitudinal, observational investigation aimed at filling the gap between controlled clinical trials and the clinical reality of medicinal cannabis use in Brazil. Under current Brazilian regulations (RDC 327/2019 and RDC 660/2022), patients access cannabinoid-based products primarily through compassionate use. This study adopts a Real-World Evidence (RWE) approach to evaluate how these treatments perform across a heterogeneous population with various comorbidities and treatment regimens.

Study Design and Procedures Participants who have already been prescribed cannabis-based products by their physicians will be recruited. The study does not interfere with medical prescriptions, dosages, or product choices.

Data collection will be conducted at three specific time points over a 180-day (6-month) period:

Baseline (T0): Collection of demographic data, medical history, primary reason for cannabis use, and previous conventional treatments. Initial scores for pain, anxiety, depression, and quality of life will be recorded.

Intermediate Follow-up (T1 - 90 days): Assessment of clinical evolution and monitoring of any early adverse events.

Final Assessment (T2 - 180 days): Final evaluation of therapeutic efficacy and overall impact on the patient's quality of life.

Instruments and Measurements To ensure objective quantification of subjective symptoms, the following validated psychometric and clinical tools will be utilized:

Quality of Life: The WHOQOL-Bref (World Health Organization Quality of Life) and EUROQOL-5D scales.

Clinical Symptomatology: The Visual Analogue Scale (VAS) for pain intensity, the Beck Depression Inventory (BDI), and the Beck Anxiety Inventory (BAI).

Safety Profile: The UKU Side Effect Rating Scale will be used to document the frequency, severity, and nature of adverse drug reactions (ADRs).

Data Management and Analysis Data will be collected via secure digital platforms (Google Forms/WhatsApp). Statistical analysis will include descriptive statistics for demographic characterization and inferential analysis (e.g., paired t-tests or non-parametric equivalents) to compare baseline scores against the 3-month and 6-month follow-ups. The study intends to identify patterns of efficacy based on the cannabinoid profile (CBD-dominant, THC-dominant, or balanced) and the specific medical conditions treated.

Ethical Compliance The study is conducted in accordance with the Declaration of Helsinki and submitted for approval by the Research Ethics Committee of the Federal University of Santa Catarina (CEP/UFSC). All participants must provide electronic Informed Consent (ICF) before data collection begins.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Residents of Brazil.
* Patients who have a valid medical prescription for cannabis-based products.
* Patients who are either starting a new treatment or are already using cannabinoid products under the ANVISA RDC 660/22 or RDC 327/19 regulations.
* Capability to understand and sign the Informed Consent Form (ICF).
* Access to a smartphone or computer with internet to complete the digital follow-up questionnaires.

Exclusion Criteria:

* Patients who do not agree to the terms of the Informed Consent Form (ICF).
* Patients who fail to complete the initial (Baseline/T0) sociodemographic and clinical questionnaires.
* Inability to communicate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study targets a diverse population of patients in Brazil who seek cannabinoid therapy for various medical conditions, primarily chronic pain, anxiety, and depression, through the pharmaceutical and clinical service flow of partner companies and clinics.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life Scores | Baseline, 45 days, 75 days, 105 days, 135 days, and 180 days.
  Evaluation of the patient's quality of life using the WHOQOL-Bref questionnaire (World Health Organization Quality of Life). This scale evaluates physical, psychological, social relationships, and environment domains. Scores range from 0 to 100, where higher scores indicate a better quality of life.

SECONDARY OUTCOMES:
Change in Pain Intensity | Baseline, 45 days, 75 days, 105 days, 135 days, and 180 days.
  Assessment of pain using the Visual Analogue Scale (VAS). Patients report their pain level on a scale from 0 (no pain) to 10 (worst possible pain).
Change in Depression Severity | Baseline, 45 days, 75 days, 105 days, 135 days, and 180 days.
  Measured by the Beck Depression Inventory (BDI). It consists of 21 items. Total scores range from 0 to 63, with higher scores indicating increased severity of depressive symptoms.
Change in Anxiety Severity | Baseline, 45 days, 75 days, 105 days, 135 days, and 180 days.
  Measured by the Beck Anxiety Inventory (BAI). It consists of 21 items. Total scores range from 0 to 63, with higher scores indicating more severe anxiety symptoms.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From Day 45 through Month 6.
  Evaluation of side effects using the UKU Side Effect Rating Scale. This scale monitors psychic, neurological, autonomic, and other side effects. It will be used to document the safety profile of the cannabinoid products.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Santa Catarina (UFSC), Centro de Ciências Biológicas (CCB), Campus Universitário, Trindade, Florianópolis - SC., Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected during the study will be shared in a de-identified format.
  Data access will be granted to researchers whose proposed use of the data has been formally approved by an independent review committee.
  The sharing process strictly complies with the Brazilian General Data Protection Law (LGPD).
  De-identified raw data concerning quality of life scores obtained through WHOQOL-Bref and EUROQOL-5D instruments. Clinical evolution scores for pain (Visual Analogue Scale - VAS), anxiety (Beck Anxiety Inventory - BAI), and depression (Beck Depression Inventory - BDI). Reported adverse events collected via the UKU Side Effect Rating Scale.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting 6 months after the publication of the final study results.
  Data availability will end 36 months after publication.
Access Criteria: Data will be shared through a secure file transfer or via the Zenodo repository using the de-identification standards already planned to ensure participant confidentiality.

REFERENCES:
- [Background] Pertwee RG. The diverse CB1 and CB2 receptor pharmacology of three plant cannabinoids: delta9-tetrahydrocannabinol, cannabidiol and delta9-tetrahydrocannabivarin. Br J Pharmacol. 2008 Jan;153(2):199-215. doi: 10.1038/sj.bjp.0707442. Epub 2007 Sep 10. PMID 17828291
- [Background] Cristino L, Bisogno T, Di Marzo V. Cannabinoids and the expanded endocannabinoid system in neurological disorders. Nat Rev Neurol. 2020 Jan;16(1):9-29. doi: 10.1038/s41582-019-0284-z. Epub 2019 Dec 12. PMID 31831863
- [Background] Maccarrone M, Di Marzo V, Gertsch J, Grether U, Howlett AC, Hua T, Makriyannis A, Piomelli D, Ueda N, van der Stelt M. Goods and Bads of the Endocannabinoid System as a Therapeutic Target: Lessons Learned after 30 Years. Pharmacol Rev. 2023 Sep;75(5):885-958. doi: 10.1124/pharmrev.122.000600. Epub 2023 May 10. PMID 37164640
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] Bhatt A. Conducting real-world evidence studies in India. Perspect Clin Res. 2019 Apr-Jun;10(2):51-56. doi: 10.4103/picr.PICR_8_19. PMID 31008069
- [Background] Kim HS, Lee S, Kim JH. Real-world Evidence versus Randomized Controlled Trial: Clinical Research Based on Electronic Medical Records. J Korean Med Sci. 2018 Jun 26;33(34):e213. doi: 10.3346/jkms.2018.33.e213. eCollection 2018 Aug 20. PMID 30127705
- [Background] Chodankar D. Introduction to real-world evidence studies. Perspect Clin Res. 2021 Jul-Sep;12(3):171-174. doi: 10.4103/picr.picr_62_21. Epub 2021 Jul 7. No abstract available. PMID 34386383